CLINICAL TRIAL: NCT06654297
Title: The Safety and Feasibility of Neoadjuvant Camrelizumab With Palbociclib for the Treatment of Resectable Esophageal Squamous Cell Carcinoma：A Phase 1 Trial
Brief Title: Neoadjuvant Camrelizumab With Palbociclib for Resectable Esophageal Squamous Cell Carcinomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, Sichuan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1551-E
Record Dates: First submitted 2024-07-20; First posted 2024-10-23 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camrelizumab+Palbociclib(100mg) 3 patients (Experimental): For palbociclib, there is 2 dose levels, 100mg qd and 125 mg qd, and if no patients experience DLT on 100mg level, 125mg level will be administered.
  Interventions: Drug: Camrelizumab; Drug: Palbociclib(100mg)
- Camrelizumab+Palbociclib(125mg) 3 patients (Experimental): For palbociclib, there is 2 dose levels, 100mg qd and 125 mg qd, and if no patients experience DLT on 100mg level, 125mg level will be administered.
  Interventions: Drug: Camrelizumab; Drug: Palbociclib(125mg)

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab will be given at at a dose of 200 mg intravenously on day 23 of a planned 28-day cycle, and two doses before surgery.
Drug: Palbociclib(100mg) — Palbociclib will be given at a dose of 100 mg every day orally with three weeks on and one week off. Four weeks is a cycle and it will be given for three cycles.
  Arms: Camrelizumab+Palbociclib(100mg) 3 patients
Drug: Palbociclib(125mg) — Palbociclib will be given at a dose of 125 mg every day orally with three weeks on and one week off. Four weeks is a cycle and it will be given for three cycles.
  Arms: Camrelizumab+Palbociclib(125mg) 3 patients

SUMMARY:
The purpose of this study is to explore the safety and feasibility of anti-programmed cell death 1(PD-1) immunotherapy, Camrelizumab, combined with cyclin-dependent kinase 4/6 blockade, Palbociclib, as a new neoadjuvant treatment regimen for patients with resectable esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with esophageal squamous cell cancer by gastroscopic biopsies.
* The primary tumor should be located in the thorax and evaluated resectable( cT1b-T3N1-3M0, cT3N0M0) by CT/MRI/EUS
* The patients should be at the range of 18-75 years old, Eastern Cooperative Oncology Group (ECOG) 0-1.
* The patients should have no functional disorders in major organs. Blood routine tests, as well as lung, liver, kidney, and heart functions should be basically normal.
* The patients should be able to understand our research and be willing to accept surgical treatment and sign the informed consent.

Exclusion Criteria:

* The stage of tumor is T4b (AJCC/International Union Against Cancer (UICC) 8th Edition) and cannot be resected.
* Currently undergoing other chemotherapy, radiotherapy, targeted therapy or immunotherapy.
* History of other malignancies.
* Have an active autoimmune disease requiring systemic treatment or a documented history of clinically severe autoimmune disease.
* Any history of allergic disease, or a sever hypersensitivity reaction to drugs, or allergy to the study drug components.
* Presence of serious medical diseases, such as grade II and above cardiac dysfunction (NYHA criteria), ischemic heart diseases, etc.
* The patients with severe systematic intercurrent diseases, including active infection or poorly controlled diabetes, coagulation disorders, hemorrhagic tendency, or those undergoing thrombolysis or anticoagulant therapy etc. are excluded from the study.
* Female participants who test positive for a serum pregnancy test, are in the lactation period, or are at a childbearing stage and unwilling to use contraception measures during the research are excluded.
* Received any investigational drug within 4 weeks prior to the first dose, or concurrently enrolled in another clinical trial.
* Any other factors that are not suitable for inclusion in this study judged by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-08-04 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Safety of combination camrelizumab and palbociclib as assessed by number of participants who experience adverse events | up to 15 weeks
  Number of participants who experience grade 1 or higher adverse events, as defined by Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0)
Feasibility of combination camrelizumab and palbociclib as assessed by number of participants who experience adverse events | up to 15 weeks
  Patients proceed to surgery without experiencing prolonged treatment-related delays. An extended treatment-related delay will be considered if it exceeds 37 days from the initially scheduled surgery date. In terms of feasibility, if there is any treatment toxicity of any grade that could adversely impact prognosis, as judged by the investigators, the planned operative date should be re-evaluated.

SECONDARY OUTCOMES:
Maximum Tolerated Dose (MTD) of palbociclib as determined by number of participants with dose limiting toxicities (DLT) | up to 15 weeks
  Maximum tolerated dose will be determined by the maximum dose at which the least number of participants experience dose-limiting toxicity. The dose limiting toxicity is defined using the Common Terminology Criteria for Adverse Events (CTCAE).
Major Pathologic Response | up to 15 weeks
  Major Pathologic Response (MPR) was defined as fewer than 10% viable tumor cells.
Objective response rate (ORR) | up to 15 weeks
  Proportion of participants with measurable disease at baseline and have been re-evaluated after at least 1 cycle of therapy with observed reduction in tumor burden as defined by RECIST and iRECIST criteria after 2 doses of Proportion of participants with measurable disease at baseline and have been re-evaluated after at least 1 cycle of therapy with observed reduction in tumor burden as defined by RECIST and iRECIST criteria after 2 doses of camrelizumab and palbociclib
Progression free survival(PFS) | Up to 2 years
  Proportion of participants who achieve progression free survival post treatment
Overall survival (OS) | Up to 2 years
  Proportion of participants who achieve survival post treatment

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Lordick F, D'Journo XB, Cerfolio RJ, Korst RJ, Novoa NM, Swanson SJ, Brunelli A, Ismail M, Fernando HC, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J; AME Thoracic Surgery Collaborative Group. Neoadjuvant Chemoradiotherapy Followed by Surgery Versus Surgery Alone for Locally Advanced Squamous Cell Carcinoma of the Esophagus (NEOCRTEC5010): A Phase III Multicenter, Randomized, Open-Label Clinical Trial. J Clin Oncol. 2018 Sep 20;36(27):2796-2803. doi: 10.1200/JCO.2018.79.1483. Epub 2018 Aug 8. PMID 30089078
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Yang H, Liu H, Chen Y, Zhu C, Fang W, Yu Z, Mao W, Xiang J, Han Y, Chen Z, Yang H, Wang J, Pang Q, Zheng X, Yang H, Li T, Zhang X, Li Q, Wang G, Chen B, Mao T, Kong M, Guo X, Lin T, Liu M, Fu J. Long-term Efficacy of Neoadjuvant Chemoradiotherapy Plus Surgery for the Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma: The NEOCRTEC5010 Randomized Clinical Trial. JAMA Surg. 2021 Aug 1;156(8):721-729. doi: 10.1001/jamasurg.2021.2373. PMID 34160577
- [Background] Tang H, Wang H, Fang Y, Zhu JY, Yin J, Shen YX, Zeng ZC, Jiang DX, Hou YY, Du M, Lian CH, Zhao Q, Jiang HJ, Gong L, Li ZG, Liu J, Xie DY, Li WF, Chen C, Zheng B, Chen KN, Dai L, Liao YD, Li K, Li HC, Zhao NQ, Tan LJ. Neoadjuvant chemoradiotherapy versus neoadjuvant chemotherapy followed by minimally invasive esophagectomy for locally advanced esophageal squamous cell carcinoma: a prospective multicenter randomized clinical trial. Ann Oncol. 2023 Feb;34(2):163-172. doi: 10.1016/j.annonc.2022.10.508. Epub 2022 Nov 15. PMID 36400384
- [Background] Shapiro J, van Lanschot JJB, Hulshof MCCM, van Hagen P, van Berge Henegouwen MI, Wijnhoven BPL, van Laarhoven HWM, Nieuwenhuijzen GAP, Hospers GAP, Bonenkamp JJ, Cuesta MA, Blaisse RJB, Busch ORC, Ten Kate FJW, Creemers GM, Punt CJA, Plukker JTM, Verheul HMW, Bilgen EJS, van Dekken H, van der Sangen MJC, Rozema T, Biermann K, Beukema JC, Piet AHM, van Rij CM, Reinders JG, Tilanus HW, Steyerberg EW, van der Gaast A; CROSS study group. Neoadjuvant chemoradiotherapy plus surgery versus surgery alone for oesophageal or junctional cancer (CROSS): long-term results of a randomised controlled trial. Lancet Oncol. 2015 Sep;16(9):1090-1098. doi: 10.1016/S1470-2045(15)00040-6. Epub 2015 Aug 5. PMID 26254683
- [Background] Doki Y, Ajani JA, Kato K, Xu J, Wyrwicz L, Motoyama S, Ogata T, Kawakami H, Hsu CH, Adenis A, El Hajbi F, Di Bartolomeo M, Braghiroli MI, Holtved E, Ostoich SA, Kim HR, Ueno M, Mansoor W, Yang WC, Liu T, Bridgewater J, Makino T, Xynos I, Liu X, Lei M, Kondo K, Patel A, Gricar J, Chau I, Kitagawa Y; CheckMate 648 Trial Investigators. Nivolumab Combination Therapy in Advanced Esophageal Squamous-Cell Carcinoma. N Engl J Med. 2022 Feb 3;386(5):449-462. doi: 10.1056/NEJMoa2111380. PMID 35108470
- [Background] Kelly RJ, Ajani JA, Kuzdzal J, Zander T, Van Cutsem E, Piessen G, Mendez G, Feliciano J, Motoyama S, Lievre A, Uronis H, Elimova E, Grootscholten C, Geboes K, Zafar S, Snow S, Ko AH, Feeney K, Schenker M, Kocon P, Zhang J, Zhu L, Lei M, Singh P, Kondo K, Cleary JM, Moehler M; CheckMate 577 Investigators. Adjuvant Nivolumab in Resected Esophageal or Gastroesophageal Junction Cancer. N Engl J Med. 2021 Apr 1;384(13):1191-1203. doi: 10.1056/NEJMoa2032125. Erratum In: N Engl J Med. 2023 Feb 16;388(7):672. doi: 10.1056/NEJMx220014. PMID 33789008
- [Background] Yin J, Yuan J, Li Y, Fang Y, Wang R, Jiao H, Tang H, Zhang S, Lin S, Su F, Gu J, Jiang T, Lin D, Huang Z, Du C, Wu K, Tan L, Zhou Q. Neoadjuvant adebrelimab in locally advanced resectable esophageal squamous cell carcinoma: a phase 1b trial. Nat Med. 2023 Aug;29(8):2068-2078. doi: 10.1038/s41591-023-02469-3. Epub 2023 Jul 24. PMID 37488287
- [Background] Solomon B, Callejo A, Bar J, Berchem G, Bazhenova L, Saintigny P, Wunder F, Raynaud J, Girard N, Lee JJ, Sulaiman R, Prouse B, Bresson C, Ventura H, Magidi S, Rubin E, Young B, Onn A, Leyland-Jones B, Schilsky RL, Lazar V, Felip E, Kurzrock R. A WIN Consortium phase I study exploring avelumab, palbociclib, and axitinib in advanced non-small cell lung cancer. Cancer Med. 2022 Jul;11(14):2790-2800. doi: 10.1002/cam4.4635. Epub 2022 Mar 20. PMID 35307972
- [Background] Dennis MJ, Sacco AG, Qi Y, Bykowski J, Pittman E, Chen R, Messer K, Cohen EEW, Gold KA. A phase I study of avelumab, palbociclib, and cetuximab in patients with recurrent or metastatic head and neck squamous cell carcinoma. Oral Oncol. 2022 Dec;135:106219. doi: 10.1016/j.oraloncology.2022.106219. Epub 2022 Oct 21. PMID 36279618
- [Background] Mody MD, Rocco JW, Yom SS, Haddad RI, Saba NF. Head and neck cancer. Lancet. 2021 Dec 18;398(10318):2289-2299. doi: 10.1016/S0140-6736(21)01550-6. Epub 2021 Sep 22. PMID 34562395
- [Background] Vermorken JB, Mesia R, Rivera F, Remenar E, Kawecki A, Rottey S, Erfan J, Zabolotnyy D, Kienzer HR, Cupissol D, Peyrade F, Benasso M, Vynnychenko I, De Raucourt D, Bokemeyer C, Schueler A, Amellal N, Hitt R. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N Engl J Med. 2008 Sep 11;359(11):1116-27. doi: 10.1056/NEJMoa0802656. PMID 18784101
- [Background] Ferris RL, Blumenschein G Jr, Fayette J, Guigay J, Colevas AD, Licitra L, Harrington K, Kasper S, Vokes EE, Even C, Worden F, Saba NF, Iglesias Docampo LC, Haddad R, Rordorf T, Kiyota N, Tahara M, Monga M, Lynch M, Geese WJ, Kopit J, Shaw JW, Gillison ML. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck. N Engl J Med. 2016 Nov 10;375(19):1856-1867. doi: 10.1056/NEJMoa1602252. Epub 2016 Oct 8. PMID 27718784
- [Background] Saba NF, Steuer CE, Ekpenyong A, McCook-Veal A, Magliocca K, Patel M, Schmitt NC, Stokes W, Bates JE, Rudra S, Remick J, McDonald M, Abousaud M, Tan AC, Fadlullah MZH, Chaudhary R, Muzaffar J, Kirtane K, Liu Y, Chen GZ, Shin DM, Teng Y, Chung CH. Pembrolizumab and cabozantinib in recurrent metastatic head and neck squamous cell carcinoma: a phase 2 trial. Nat Med. 2023 Apr;29(4):880-887. doi: 10.1038/s41591-023-02275-x. Epub 2023 Apr 3. PMID 37012550
- [Background] Ju WT, Xia RH, Zhu DW, Dou SJ, Zhu GP, Dong MJ, Wang LZ, Sun Q, Zhao TC, Zhou ZH, Liang SY, Huang YY, Tang Y, Wu SC, Xia J, Chen SQ, Bai YZ, Li J, Zhu Q, Zhong LP. A pilot study of neoadjuvant combination of anti-PD-1 camrelizumab and VEGFR2 inhibitor apatinib for locally advanced resectable oral squamous cell carcinoma. Nat Commun. 2022 Sep 14;13(1):5378. doi: 10.1038/s41467-022-33080-8. PMID 36104359